CLINICAL TRIAL: NCT00282529
Title: Identification of a Screening Tool and Treatment of Lymphedema Secondary to the Management of Breast Cancer Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J05101
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; Lymphedema
Keywords: lymphedema, screening, treatment
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

INTERVENTIONS:
Device: High Risk Lymphedema Education and Device Intervention

SUMMARY:
The proposed research is designed to establish lymphedema incidence rates for a varied population of breast cancer patients. Patients with breast preservation, mastectomy, sentinel lymph node biopsy, axillary dissection and radiation therapy will be included with the goal of determining the impact that each of these treatments has on development of lymphedema. Establishing incidence in these populations is crucial to the remainder of the study. We conduct a two phase study. The first phase will use arm measurements, a symptom survey (The Lymphedema and Breast Questionnaire), a functional survey (Disability of the Arm, Shoulder, and Hand Questionnaire), and operative and pathology information to create a simple screening tool to predict the development of lymphedema. Currently, lymphedema is only diagnosed after arm swelling develops. The goal of the screening tool is to identify those patients at significantly increased risk for development of lymphedema as compared to the general population of breast cancer survivors. Phase 2 of the study will test a lymphedema prevention strategy in a high risk population. The goal of this phase is to reduce the incidence of lymphedema in those patients that have undergone an axillary node dissection with radiation therapy by using a combination of education, a compression sleeve and decongestive exercises. If prevention is successful, the development of a screening tool becomes even more important to identify those patients that should undergo a prevention regimen.

DETAILED DESCRIPTION:
Background: Lymphedema has varied definitions, all based on limb volume changes. None incorporates limb volume changes, symptoms, and functional deficits. We will determine the incidence of lymphedema in breast cancer patients and the impact of breast conserving therapy, radiation therapy, sentinel lymph node biopsy, and axillary node dissection. The impact of lymphedema can be evaluated in a number of ways; 1) The Lymphedema and Breast Cancer Questionnaire (LBCQ) identifies symptoms that are unique to patients with lymphedema and 2) The Disability of the Arm, Hand, and Shoulder (DASH) survey will be used to determine the functional impact of lymphedema.

Objective/Hypothesis: Our hypotheses are: 1) Local therapies for breast cancer result in different lymphedema rates depending on the combination of therapies used. 2) A simple screening tool that incorporates symptoms, limb volume measurements, and tumor staging and treatment modalities can predict those patients that will develop lymphedema. 3) Functional impairment of the arm is severe in patients with lymphedema. 4) Prevention of lymphedema in a high risk population is possible with education, a compression sleeve, and decongestive exercise.

Specific Aims: 1) Evaluate patients both pre-operatively and at specific time intervals post-operatively to establish the incidence of lymphedema in sentinel lymph node biopsy and axillary dissection groups. 2) Create a simple screening tool using arm measurements, symptoms identified by the LBCQ, and treatment and staging information to identify patients that should go on to further testing and treatment. 3) Utilize the DASH survey to measure the extent of disability from lymphedema and surgical treatment. 4) Conduct a randomized trial of lymphedema prevention in a high-risk breast cancer population.

Study Design: This proposal will be conducted in two phases. Phase 1 will accomplish Specific Aim 1, 2, and 3. Patients with newly diagnosed breast cancer awaiting definitive surgery, will be enrolled pre-operatively and undergo arm measurements and complete the LBCQ and the DASH surveys. These same study procedures will be completed at 1, 3, 6, 12, 18, and 24 months postoperative. Documentation collected during the study will include: demographic information; co-morbid conditions; operative and pathology reports; and use of adjuvant therapies such as chemotherapy, hormonal therapy, and radiation therapy. Incidence rates of lymphedema and the impact of extent of surgery and radiation therapy will be determined. We will also use this information to develop a simple screening tool to identify patients that will develop lymphedema prior to the development of significant limb volume changes. Specific Aim 4 is Phase 2 of the proposal. A high risk population (those that have an axillary node dissection and radiation therapy) will be randomized to standard education versus standard education, compression sleeve, and exercise. The effectiveness of prevention to reduce incidence and severity of lymphedema and the impact on symptoms and functional impairment will be determined. This work will move toward a new paradigm of lymphedema management with a simple screening tool to identify high risk patients before significant swelling occurs and investigate prevention strategies to decrease the incidence of lymphedema.

Cancer Relevance: Lymphedema is a feared complication of breast cancer treatment. Currently it is recognized and treated only after development of significant limb volume changes when it is symptomatic and difficult to treat. Documentation of the impact of local therapies on the development of lymphedema will allow clinicians to make more informed decisions regarding risk benefit ratios of each of our local therapies. Development of a screening tool will allow us to identify high risk populations. Ideally, the high risk population will be identified and an effective prevention strategy implemented. Phase one of this study will help to answer the questions regarding incidence and create a screening tool and phase two will allow the evaluation of a prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

Age of 18 years or older, biopsy proven breast cancer with no known metastatic cancer, surgical management of breast cancer with node evaluation to be completed at Johns Hopkins Hospital, ability to speak and read English, willing and able to continue follow-up at Johns Hopkins Avon foundation Breast Center -

Exclusion Criteria: Known psychiatric illness, unwillingness to be followed for two years, functional arm deficits, prior radiation therapy to the breast or axilla, any prior diagnosis of cancer except basal cell cancer

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-01 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Bilateral arm measurements, Lymphedema and Breast Cancer Questionnaire, Disability of the Arm and Shoulder and Hand(DASH)Questionnaire

SECONDARY OUTCOMES:
Standard lymphedema risk reduction education, Lymphedema prevention

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Jacobs, M.D., Principal Investigator — Johns Hopkins Medical Institutions, Department of Surgery
Locations (1):
- Avon Breasts Center, Johns Hopkins Medical Institutions, Baltimore, Maryland, United States